CLINICAL TRIAL: NCT02608788
Title: Comparing the Efficacies Between the Spray of S.L. Spray Solution and Difflam and Acular to Release Postoperative Sore Throat
Brief Title: S.L. Spray Solution® and Difflam® and Acular®Spray for the Prevention of Postoperative Sore Throat
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 103-2453A3
Record Dates: First submitted 2015-10-16; First posted 2015-11-20 (Estimated); Last update posted 2021-05-21 (Actual); Status verified 2015-10

CONDITIONS: Sore Throat
Keywords: postoperative sore throat; American Society of Anesthesiologists status; general anesthesia; post-anesthesia care unit(PACU)
MeSH Terms: conditions — Pharyngitis | interventions — Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- S.L.® & Difflam Forte ® (Active Comparator): "1.5 mg/ml Benzydamine" , "S.L.® Spray Solution" 2.5 mg and "3.0 mg/ml Benzydamine" ,Difflam Forte ® 5.0 mg spray by mouth. Before intubation, each endotracheal tube cuff was scattered 10 times of spray by physicians that might cover 20 cm long of the cuff.
  Interventions: Drug: S.L.®
- placebo ( for Acular® ) (Placebo Comparator): placebo(distilled water)spray by mouth. Before intubation, each endotracheal tube cuff was scattered 10 times of spray by physicians that might cover 20 cm long of the cuff.
  Interventions: Drug: placebo
- Acular® & S.L.® (Active Comparator): "5％ Ketorolac Tromethamine" , "Acular®" 8.0 mg and "1.5 mg/ml Benzydamine" , "S.L.® Spray Solution" 2.5 mg spray by mouth. Before intubation, each endotracheal tube cuff was scattered 10 times of spray by physicians that might cover 20 cm long of the cuff.
  Interventions: Drug: Acular®
- Difflam Forte ® & Acular® (Experimental): "3.0 mg/ml Benzydamine" , "Difflam Forte ®" 5.0 mg and "5％ Ketorolac Tromethamine" "Acular®" 8.0 mg spray by mouth. Before intubation, each endotracheal tube cuff was scattered 10 times of spray by physicians that might cover 20 cm long of the cuff.
  Interventions: Drug: Difflam Forte ®

INTERVENTIONS:
Drug: S.L.® — "1.5mg/ml Benzydamine hydrochloride"," S.L.®" spray by mouth . Before intubation, each endotracheal tube cuff was scattered 10 times of spray by physicians that might cover 20 cm long of the cuff.
  Other Names: Andolex®
  Arms: S.L.® & Difflam Forte ®
Drug: Difflam Forte ® — "3.0mg/ml Benzydamine hydrochloride" , " Difflam Forte ®" spray by mouth . Before intubation, each endotracheal tube cuff was scattered 10 times of spray by physicians that might cover 20 cm long of the cuff.
  Other Names: Tantum Verde®
  Arms: Difflam Forte ® & Acular®
Drug: Acular® — "5％ Ketorolac Tromethamine" , " Acular® " spray by mouth . Before intubation, each endotracheal tube cuff was scattered 10 times of spray by physicians that might cover 20 cm long of the cuff.
  Other Names: Apo-Ketorolac® Ophthalmic
  Arms: Acular® & S.L.®
Drug: placebo — Distilled water spray by mouth. Before intubation, each endotracheal tube cuff was scattered 10 times of spray by physicians that might cover 20 cm long of the cuff.
  Other Names: distilled water
  Arms: placebo ( for Acular® )

SUMMARY:
The purpose of intubation for patients under general anesthesia is to maintain their respiratory function. However, this procedure does cause a postoperative sore throat. Comfort of patients could be promoted if effective treatment could be found.

The specific aims of this project are:

1. Comparing the Efficacies Between the Spray of S.L. Spray Solution and Difflam to Release Postoperative Sore Throat.
2. Acular spray for the prevention of postoperative sore throat.
3. Comparing the Efficacies Between the Spray of S.L. Spray Solution and Difflam and Acular to Release Postoperative Sore Throat.

DETAILED DESCRIPTION:
This is a quasi-experimental study with purposive sampling. Patients were distributed into the four groups (1.5mg / ml Benzydamine hydrochloride, 3.0mg / ml Benzydamine hydrochloride, 5％Ketorolac Tromethamine) by the operative room. Research tools including pain scale (Numeric Rating Scale: 0-10), drugs and case data record sheet. Collected information was managed by SPSS for Windows (version 21.0) statistical software package. Both the descriptive and Inferential statistics were performed. Sample homogeneity among the four groups were verified by F-test and chi-square test. generalized estimating equation was selected to compare the throat pain in the four points of assessment.

The specific aims of this project are:

1. Comparing the Efficacies Between the Spray of S.L. Spray Solution and Difflam to Release Postoperative Sore Throat.
2. Acular spray for the prevention of postoperative sore throat.
3. Comparing the Efficacies Between the Spray of S.L. Spray Solution and Difflam and Acular to Release Postoperative Sore Throat.

ELIGIBILITY:
Inclusion Criteria:

1. intubation for patients under general anesthesia
2. age>20
3. none pre-operative sore throat
4. by the researchers explain research purposes, the researchers agreed to participate

Exclusion Criteria:

1. postoperative on N-G tube
2. Surgical side is located by the mouth or throat
3. thyroidectomy
4. difficult airway
5. none extubation at PACU
6. on patient-controlled analgesia
7. the medical records have a history of nonsteroidal antiinflammatory drugs allergy
8. medical records have kidney disease or a history of renal dysfunction
9. peptic ulcer
10. pregnancy or lactation

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2014-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
pain scale (Numeric Rating Scale: 0-10) | 1.5 year

SECONDARY OUTCOMES:
nonsteroidal antiinflammatory drug side effect | 1.5 year

CONTACTS AND LOCATIONS:
Overall Officials: Hsiu-Ling Yang, RN, MS, Principal Investigator — Chang Gung Memorial Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hung NK, Wu CT, Chan SM, Lu CH, Huang YS, Yeh CC, Lee MS, Cherng CH. Effect on postoperative sore throat of spraying the endotracheal tube cuff with benzydamine hydrochloride, 10% lidocaine, and 2% lidocaine. Anesth Analg. 2010 Oct;111(4):882-6. doi: 10.1213/ANE.0b013e3181d4854e. Epub 2010 Mar 19. PMID 20304980